CLINICAL TRIAL: NCT05609292
Title: Testing A Visual Thermometer in Newborns and Young Infants
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: new
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hyperthermia; Hypothermia
Keywords: temperature monitoring; liquid crystal thermometer; hypothermia; hyperthermia; LCTD; infant temperature; infant hyperthermia; infant hypothermia; neonate hyperthermia; neonate hypothermia; neonate temperature
MeSH Terms: conditions — Hyperthermia; Hypothermia | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Infants will get their temperature measured with the liquid crystal thermometer. We are not providing any interventions as they will be in the care of a healthcare team.
  Interventions: Device: observational

INTERVENTIONS:
Device: observational — Infants will get their temperature measured with the liquid crystal thermometer. We are not providing any interventions as they will be in the care of a healthcare team.

SUMMARY:
"Severe neonatal jaundice and acute bilirubin encephalopathy are a major cause of death and disability among newborns in LMICs. Filtered sunlight phototherapy (FSPT) was developed, tested and shown to be safe and efficacious in the treatment of jaundice, because effective electric-powered conventional phototherapy is often unavailable10,11. However, FSPT currently requires at least hourly temperature monitoring by healthcare providers (HCPs) because infants receiving FSPT are prone to both hypothermia and hyperthermia.

20 years ago, a liquid crystal thermometer, ThermospotTM (Maternova, Providence, RI) was developed primarily for use in LMICs. It was designed to detect hypothermia and is most sensitive in cold infants and not as sensitive as needed for detecting hyperthermia or fever. The purpose of this pilot study is to determine the accuracy and useability of this LCTD for a wider spectrum of temperatures when used in a large group of infants in a high-income country. If the device performs well in this study, we plan to study it in a low- and middle-income country in Africa."

ELIGIBILITY:
Inclusion Criteria:

* Infants 0-6 months (<7 months) presenting to Masonic Emergency Room or inpatient ward, their parent or caregiver who provide verbal consent in English or through a medical interpreter.

Exclusion Criteria:

* Any infant undergoing active resuscitation
* any infant for whom physician deems study enrollment would interfere with their care
* any infant whose parents or caregiver decline enrollment
* any nurse or other healthcare provider who declines participation
* Parents who do not understand English, and do not have a medical interpreter at the bedside.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants between the age of 0-6months
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of the liquid crystal thermometer with measuring a temperature | baseline
  determining the accuracy of the LCTD in estimating the temperature of infants 0-6 months presenting to the emergency room for treatment
Parents/Caregivers and Healthcare provider accuracy in evaluating the infant temperature | baseline
  Our secondary endpoint is determining parents/caregivers and healthcare provider accuracy in evaluating the temperature of their infant or the infant they are caring for and determining the category of the temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Slusher, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No